CLINICAL TRIAL: NCT03710993
Title: Beddr Sleep SpO2 Equivalency Calibration Study
Brief Title: Accuracy Assessment of Beddr Oximeter
Status: Completed | Type: Observational
Sponsor: Hancock Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR 2018-290
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Oximetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: oximeter — Participants breathe a controlled gas mixture to induce several reduced oxygen states while oximeter measurements are taken for comparison to corresponding transfer standard and reference devices to assess oximeter calibration and accuracy.

SUMMARY:
Accuracy performance of Beddr oximeter

DETAILED DESCRIPTION:
This study will evaluate the accuracy of the Beddr sleepTuner oximeter compared to a transfer standard and multiple reference devices.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Adult subjects 18 up to 50 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker or who has not smoked within 2 days prior to the study.
* Male or female of any race
* Subject demographics include a range of skin pigmentations, including at least 1 darkly pigmented subjects or 15% of the subject pool, whichever is larger.

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Females who are pregnant, who are trying to get pregnant or who have a urine test positive for pregnancy on the day of the study
* Subjects with known respiratory conditions such as:

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * unresolved respiratory or lung surgery with continued indications of health issues,
  * emphysema, COPD, lung disease
* Subjects with known heart or cardiovascular conditions such as:

  * Hypertension: systolic >140mmHg, Diastolic >90mmHg on 3 consecutive readings.
  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury within the last 2 months,
  * cancer / chemotherapy
* Subjects with known clotting disorders

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
* Subjects with Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
* Unwillingness or inability to remove colored nail polish or non-clear artificial nails from test digits.
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers, ranging in pigmentation from light to dark.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
SpO2 accuracy | 60 minutes
  Collect and analyze data to assess SpO2 calibration and accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No